CLINICAL TRIAL: NCT02015936
Title: Physical Activity for Advanced Stage Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-17389
Record Dates: First submitted 2013-12-13; First posted 2013-12-19 (Estimated); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Cancer
Keywords: stage III cancer; stage IV cancer; cancer; advanced stage cancer; Nintendo Wii training; exercise; physical training; physical function; physical fitness test
MeSH Terms: conditions — Neoplasms; Motor Activity | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prescriped Physical Activity (Experimental): Physical fitness evaluation followed by prescribed physical activity and progress reporting.
  Interventions: Behavioral: Six Week Physical Activity Intervention; Other: Progress Reporting

INTERVENTIONS:
Behavioral: Six Week Physical Activity Intervention — Tailored Wii Fit prescription based on physical fitness assessments and a schedule of six home visits by an oncology RN.
Other: Progress Reporting — Participants will keep a log to record the physical activities they have done with the Wii Fit during the 6-week period. Audio-recording may be included for quality control. Self-report data will be collected by Internet surveys through the University of South Florida (USF) Health Qualtrics application at baseline (T1) and at 6 weeks post-intervention (T2). The nurse will take small amount of the participant's hair (20 strands) for a hormone test during the first visit and last visit.
  Other Names: documentation; self-reporting; questionnaire

SUMMARY:
The purpose of this study is to understand if a home-based physical activity program can improve symptoms and physical function among patients with advanced stage cancer.

DETAILED DESCRIPTION:
This program includes use of the Nintendo Wii Fit™Plus (Wii Fit) and home visits by a nurse. The same nurse will attend all of the visits.

ELIGIBILITY:
Inclusion Criteria:

* have stage III or IV cancer diagnosis
* able to understand English
* have a Karnofsky Performance Status (KPS) score of 60% (able to care for most of the personal needs)
* have fatigue and/or two other target symptoms
* have been cleared by their provider to engage low to moderate intensity physical activities

Exclusion Criteria:

* are hospitalized
* have lesion or metastasis of bone
* have a cardiac pacemaker
* have a history of seizure or loss of consciousness
* have been using a Wii Fit
* diagnosed cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-12-12 (Actual); Primary Completion 2015-09-14 (Actual); Study Completion 2021-10-21 (Actual)

PRIMARY OUTCOMES:
Rate of Participation Among Eligible Patients | 6 weeks per participant
  Feasibility and acceptability of a tailored Wii Fit intervention. Hypothesis1.1: 60% of eligible patients will enroll; 1.2: 60% of participants will adhere to their tailored physical activity prescriptions; 1.3: 70% of participants will agree that Wii Fit is easy to use, enjoyable, convenient, and helpful.
  Enrollment rate: ratio of number of advanced stage cancer patients enrolled in the study to total number of patients meeting eligibility criteria invited to participate in the study. Adherence rate: ratio of the number of participants who adhere to the tailored Wii Fit prescription (i.e., expend at least 60% of prescribed kilocalories each week) to the total number of participants in the study. Acceptability of and satisfaction with the intervention: ratio of number of participants whose mean scores of Wii Fit and RN Visiting Surveys are equal to or more than 3 on 1-4 Likert-type scale to the total number of participants in the study.

SECONDARY OUTCOMES:
Rate of Positive Response to Participation | 6 weeks per participant
  Examine changes in outcomes (fatigue, pain, depression, anxiety, sleep quality, physical function, perceived stress, and chronic Hypothalamus-Pituitary-Adrenal (HPA) activation) over 6 weeks among patients who have the intervention. Hypothesis 2.1: There will be positive changes in the outcomes.
  Repeated measures ANOVA will be used to compare T1 with T2 scores in fatigue, pain, depression, anxiety, sleep quality, physical function, perceived stress, and hair cortisol. Twenty participants will provide 80% power to detect only large effect sizes (d>.60), which cannot be anticipated. Because the purposes of this study are to inform future larger studies, the ANOVA will be used to calculate effect sizes (η2) for future power estimations. Because effect size calculation will be the central purpose of the ANOVAs, no adjustment will be made to reduce the possibility of Type 1 errors (p<.05).

CONTACTS AND LOCATIONS:
Overall Officials: Hsiao-Lan Wang, Ph.D., RN, Principal Investigator — University of South Florida
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States